CLINICAL TRIAL: NCT00476801
Title: The Effectiveness Of UVA1 Irradiation In The Treatment Of Skin Conditions With Altered Dermal Matrix: A Controlled, Cross-Over Study
Brief Title: UVA1 Light for Treatment of Scleroderma and Similar Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Sewon Kang, MD, Professor and Director Clinical Pharmacology, University of Michigan Department of Dermatology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Derm 438
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Scleroderma; Keloids; Other Fibrosing Conditions
Keywords: UVA1; scleroderma; keloids; light therapy; morphea
MeSH Terms: conditions — Scleroderma, Diffuse; Keloid; Scleroderma, Localized

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UVA1 irradiation (Experimental): The dose and scheduling will be similar to those being successfully used in Germany: up to 130J/cm2 from a UVA1 Sellamed irradiation device (German manufactured UVA1 light emitting device) with irradiations up to 5 times per week for up to 14 weeks on one side of the face. Then a cross-over treatment an equal length of time.
  Interventions: Device: German manufactured UVA1 light emitting device
- Control (No Intervention): No treatment on the opposite side of the face as the UVA1 treatment for up to 14 weeks. Then a cross-over treatment an equal length of time.

INTERVENTIONS:
Device: German manufactured UVA1 light emitting device — The UVA1 dose will be up to 130 J/cm2.
  Arms: UVA1 irradiation

SUMMARY:
The purpose of this investigation is to evaluate the effectiveness of an investigational device which is similar in appearance to a "tanning bed" but which emits ultraviolet irradiation of a specific wavelength known as UVA1. This device has not been approved by the FDA for general use in this country, as yet, but it has been used quite successfully in Europe for several years in treating such conditions as scleroderma, keloids, and other fibrosing conditions of the skin. Your participation in this study may yield important information regarding the safety and effectiveness of this form of light therapy for the treatment of these skin conditions which, at present, are difficult to treat.

DETAILED DESCRIPTION:
Ultraviolet rays from the sun that reach the earth surface are divided into shorter wavelength, hence high energy, UVB (290-320nm) and longer wavelength, hence low energy UVA (320-400nm). The wavelengths of light that cause sunburn and are associated with skin cancer causation is the high energy UVB. UVA wavelengths can be further divided into relatively shorter wavelength, hence higher energy UVA2 (320-340nm) and longer wavelength, lower energy UVA1 (340-400nm). Phototherapy light boxes used in our clinic for the treatment of psoriasis, atopic dermatitis, and pruritus, as well as those used in tanning salons emit both UVB and UVA wavelengths of light. The advantages of using UVA1 light source in the treatment of skin conditions are 1) lack of skin cancer and sunburn causing rays (UVB/UVA2) and 2) as a consequence, the ability to treat patients more safely.

Keloid, scleroderma, acne keloidalis nuchae, and burn scars are all characterized by collagenous thickening of the skin resulting in superficial and deep cutaneous sclerosis. Treatments for these disabling conditions are inadequate at present. Recently, in non-controlled studies, UVA1 was shown to induce improvement in patients with scleroderma, granuloma annulare and urticaria pigmentosa (1-3). The mode of action of UVA1 treatment is not completely understood, however, local immuno-modulation appears to be important (4). UVA1 has also been shown to stimulate collagenase activity in a dose dependent manner in the dermis (5,6). We postulate, therefore, that UVA1 in appropriate doses can improve these fibrosing skin conditions safely through collagenase-mediated removal of excess dermal collagen.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-80 years
* Clinical diagnosis of keloid (or hypertrophic scar), scleroderma, acne keloidalis nuchae, old burn scars, granuloma annulare, and other related conditions associated with altered dermal matrix.
* At least two areas of comparable thickness/induration, one on each side, or one large sclerotic lesion that can be divided in half for UVA1 and sham UV therapy.
* No disease states or physical conditions which would impair evaluation of the test site.
* Willing and able to receive UVA1 as directed in the protocol, make evaluation visits, and follow protocol restrictions.
* Signed, written, witnessed, informed consent form.
* Must live within driving distance of Ann Arbor, Michigan.

Exclusion Criteria:

* History of photosensitivity.
* UVA1 irradiation hypersensitivity in a UVA1 photo-provocation test.
* Pregnant or nursing women.
* Involved in an investigational study within the previous 4 weeks.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-07; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Plaque thickness, plaque hardness, patient mobility | 28 weeks

SECONDARY OUTCOMES:
Levels of collagen and mmp induction | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sewon Kang, MD, Principal Investigator — University of Michigan hospital
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States